CLINICAL TRIAL: NCT04072211
Title: Demonstration Project on Health Care Worker Protection Against Hepatitis B in Kalulushi District
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 003-01-19
Record Dates: First submitted 2019-05-22; First posted 2019-08-28 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis B Virus; Health Care Associated Infection
Keywords: Hepatitis B Virus; Vaccination; Health Personnel
MeSH Terms: conditions — Hepatitis B; Cross Infection | interventions — Engerix-B

STUDY DESIGN:
Intervention Model Description: All study participants will be screened for Hepatitis B Virus and those eligible for vaccination will receive the vaccine. Those already infected will be linked to care and those with a protective level of anti-HBs will not receive the vaccine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vaccine arm (Other): Engerix-B vaccine will be administered. This arm will include all those at risk of hepatitis B virus infection
  Interventions: Biological: Engerix-B

INTERVENTIONS:
Biological: Engerix-B — Hepatitis B vaccine administered through intramuscular injection at 0, 1, and 6 months

SUMMARY:
Hepatitis B virus (HBV) has infected over one third of the world's population; of these about 350 million go on to be chronic carriers. Infection with HBV can be self-limiting depending on age and immunity status of the infected person. Acute infection with HBV is cleared within six months of initial infection while chronic infection can last longer than six months. HBV can be transmitted perinatally, sexually, horizontally, through direct contact with infectious body fluids or blood, being pricked with an infected needle and injury from instruments contaminated with infectious body fluid or blood. Certain population groups are at higher risk of infection with HBV. Among these populations is that of health care workers (HCWs). In this population, HBV infection can occur through occupational exposure. In fact, the hepatitis B virus is more contagious than human immunodeficiency virus (HIV) during a needle stick injury (30% versus 0.5%). It is therefore imperative that HCWs are highly knowledgeable about HBV and how they can prevent transmission. Protection from HBV infection can be achieved by means of vaccination after which the HBV vaccine has been shown to be 90-100% effective.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) has infected over one third of the world's population; of these about 350 million go on to be chronic carriers. In adults, infection with HBV can be self-limiting in up to 95% of those infected and the most common route of infection is sexual transmission. HBV can also be transmitted perinatally, horizontally, through direct contact with infectious body fluids or blood, being pricked with an infected needle and injury from instruments contaminated with infectious body fluid or blood.

Certain population groups are at higher risk of infection with HBV. Among these populations is that of health care workers (HCW). In this population, HBV infection can occur through occupational exposure. It is therefore imperative that HCWs are highly knowledgeable about HBV and how they can prevent transmission.Protection from HBV infection can be achieved by means of vaccination after which the HBV vaccine has been shown to be 90-100% effective.

Despite availability of these vaccines, studies have shown low rates of vaccination against HBV amongst HCW in different countries. However, in countries where there is a deliberate policy to vaccinate HCW, the rates of HBV vaccination are over 90%. In Zambia, this rate has been reported to be as low as 19.3%.

This project will demonstrate an approach to reduce HCW risk of HBV through increasing knowledge and awareness of HBV among HCWs, providing vaccination to HCWs and linking those already carrying HBV infection to care and treatment. The study will also investigate the cost of vaccinating HCWs against HBV and evaluate feasibility, acceptability and implementation factors to inform possible scale-up of this approach throughout Zambia.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Willing to consent and meet project requirements for training and follow-up.

Exclusion Criteria:

* Kidney disease or renal failure
* Pregnant
* History or current neurological condition
* Express refusal to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Demonstrate attainment of protective Hepatitis B surface antibody (anti-HBs) levels in their serum | Eight Months
  anti-HBs will be measured at enrollment before any vaccine is administered, at one months post first, before administering the third dose, and one month post last vaccine doses.

SECONDARY OUTCOMES:
Demonstration of attained cell-mediated protection against Hepatitis B surface Antigen after vaccination. | Eight Months
  2.0×106 cells/mL will be stimulated with artificial Hepatitis B surface Antigen antigen and characterised into naïve B and T cells, effector B and T cells and memory B and T cells. This will be done by targeting specific cell surface markers using fluorochrome labelled antibodies such as anti-CD4+-ECD, CD8+-PeCy7, CD3-APC-H7, CD45RA-FITC, CD45RO-PCy7, FoxP3+-PE, CD27-PCy5, CCR7-FITC, CD20-APC, CD40-FITC, CD78-FITC, CD30-PE, CD38-PerCP-Cy5.5, CD19-PE-Cy7 and IgM-FITC. Before the cells are labelled, they will be stained and blocked using FcR blocking reagents.
Linkage of health care workers with chronic Hepatitis B virus infection to treatment and management | One Month
  Health care workers who are Hepatitis B surface Antigen positive linked to routine care
Cost and cost-effectiveness analysis of a universal Hepatitis B Virus vaccination strategy targeted at healthcare workers in Kalulushi district | Eighteen months
  The descriptive costing study will estimate the costs of a vaccination program. Assuming a bottom-up, ingredients-based approach, costs will be collected in local currency units and converted to United States Dollar (US$) using the midpoint exchange rate at the time of implementing the study. The cost-effectiveness analysis will be carried out from societal and payer's perspective.

CONTACTS AND LOCATIONS:
Locations (1):
- Kalulushi district all facilities, Kalulushi, Copperbelt, Zambia